CLINICAL TRIAL: NCT02570503
Title: Do Intraoperative Periarticular Injections Improve Postoperative Pain Control in Patients Receiving Duramorph (Preservative Free) During Total Knee Arthroplasty? A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Postoperative Pain Control After Periarticular Injection During Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study's primary aims are no longer clinically impactful, as intrathecal morphine has fallen out of favor and replaced with different agents so that outpatient/23 hr surgery is more predictably achievable.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20004125
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine; Ketorolac; Clonidine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROP/KET/CLON/EPI/SAL (Experimental): Ropivacaine (ROP) (5mg/ml)- 50ml Ketorolac (KET) (30mg/ml)- 1ml Clonidine (CLON) (0.1mg/ml)- 0.8ml Epinephrine (EPI) (1mg/ml)- 0.5ml 0.9% sodium chloride SAL)--47.7 ml
  Interventions: Drug: Ropivacaine; Drug: Ketorolac; Drug: Clonidine; Drug: Epinephrine; Drug: 0.9% sodium chloride
- Placebo (Placebo Comparator): 0.9% Sodium Chloride- 100ml
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine (5mg/ml)-50ml
  Other Names: periarticular injection
  Arms: ROP/KET/CLON/EPI/SAL
Drug: Ketorolac — ketorolac (30mg/ml)- 1 ml
  Other Names: periarticular injection
  Arms: ROP/KET/CLON/EPI/SAL
Drug: Clonidine — clonidine (0.1mg/ml)- 0.8ml
  Other Names: periarticular injection
  Arms: ROP/KET/CLON/EPI/SAL
Drug: Epinephrine — epinephrine (1mg/ml)-1ml
  Other Names: periarticular injection
  Arms: ROP/KET/CLON/EPI/SAL
Drug: 0.9% sodium chloride — Sodium chloride 0.9%- 47.7 ml
  Other Names: periarticular injection

SUMMARY:
This study will evaluate the use of a local injection around the knee (periarticular) during total knee replacement (TKR) surgery to see if it reduces postoperative pain levels. The injection is a combination of various medications which are thought to reduce pain levels.

Approximately 128 patients will participate in this study, half of the patients will receive this injection during surgery and the other half will receive a saline (salt water) injection. Pain scores after the surgery will be compared between the two groups.

All patients will also receive a long-acting (24 hours) morphine injection during surgery.

The hypothesis is that those participants receiving intrathecal Duramorph and local periarticular injections will have improved pain scores and reduced narcotic use when compared with intrathecal Duramorph alone at 48 hours postoperatively.

DETAILED DESCRIPTION:
Data Collection:

Data will be collected from the patient's medical record after discharge

Variables include:

* Age
* Sex
* BMI
* UPAT score (Universal Pain Assessment Tool)- this is assessed hourly postoperatively by nursing staff on Orthopedics Unit
* Patient's assessment of acceptability of pain
* UPAT score as assessed by physical therapy pre and post therapy sessions
* Duramorph dose
* Time patient arrived on the Orthopedic Unit
* Length of ambulation during physical therapy sessions
* Amount of supplementary opioids (measured in morphine equivalents)
* Use of anti-emetics
* Any complications of surgery including venous thromboembolic event, cardiac event, bleeding event
* Length of hospital stay

The pharmacist will randomize patients to either study arm, prepare the injection and maintain dispensing records.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Written informed consent

Exclusion Criteria:

* Pregnant women
* Creatinine clearance less than 60 ml/min
* BMI greater than 40
* Currently use greater than 80mg morphine-equivalents daily (pre-operatively)
* Receive a unicondylar knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10; Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Golladay, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Started | 34 | 30
Completed | 34 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (8.1) | 64.1 (9.4) | 64.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 19 | 14 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Universal Pain Assessment Tool (UPAT)
Description: Patient's pain scores will be measured with the UPAT scale which ranges from 0 (no pain) to 10 (severe pain) This is measured hourly while the patient is awake after the surgery.
Time Frame: 3 days after surgery
Population: Protocol was amended early in the study to omit this outcome due to apparent data irregularities - no data was collected and no outcomes can be reported
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Narcotic Use During Hospitalization
Description: The amount of narcotic pain medication needed for patient to be comfortable. This is measured in morphine equivalents since there are many pain medications other than morphine.
Time Frame: 0-24 hours post surgery period, 24 - 48 hours post surgery period, and Full 48 hours post surgery period
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Number analyzed (Participants) | 34 | 30
mg morphine equivalents
  0 to 24 hour post surgery period | 58.9 (41.2) | 72.3 (49.4)
  24 to 48 hour post surgery period | 66.5 (51.3) | 72.8 (61.7)
  Full 48 hour post surgery period | 125.6 (80.7) | 145.7 (99.2)

3. Secondary Outcome: Patient's Subjective Rating of Pain
Description: Patients are asked if their pain is acceptable (yes/no)
Time Frame: 3 days after surgery
Population: as for outcome 1
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: UPAT Score Before and After Physical Therapy
Description: Pain in score change after physical therapy
Time Frame: 3 days after surgery
Population: as for outcome 1
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Ambulation During Physical Therapy
Description: The length (in feet) patient is able to ambulate during physical therapy
Time Frame: 48 hours after surgery
Population: as for outcome 1
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 hours post surgery
Arm/Group | ROP/KET/CLON/EPI/SAL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 0/34 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02570503/Prot_SAP_000.pdf